CLINICAL TRIAL: NCT00796913
Title: Prospective Randomized Study of Therapy Withdrawal vs Continued Low Dose Medical Therapy in Patients With Graves' Disease Entering Remission During ATD Therapy
Brief Title: Remission Induction and Sustenance in Graves' Disease 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Scott Karmisholt, MD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RISG2
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Graves Disease; Hyperthyroidism
MeSH Terms: conditions — Graves Disease; Hyperthyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stop of medication after remission (Active Comparator): After enetering remission patients are randomised to continue low dose medication or to stop medication: Overview of study described in:
  Laurberg P, Nygaard B, Andersen S, Carlé A, Karmisholt J, Krejbjerg A, Pedersen IB, Andersen SL. Association between TSH-Receptor Autoimmunity, Hyperthyroidism, Goitre, and Orbitopathy in 208 Patients Included in the Remission Induction and Sustenance in Graves' Disease Study. J Thyroid Res. 2014;2014:165487. doi: 10.1155/2014/165487.
  Interventions: Other: Stop medication
- Medication for 2 yrs after remission (No Intervention): See Laurberg P, Nygaard B, Andersen S, Carlé A, Karmisholt J, Krejbjerg A, Pedersen IB, Andersen SL. Association between TSH-Receptor Autoimmunity, Hyperthyroidism, Goitre, and Orbitopathy in 208 Patients Included in the Remission Induction and Sustenance in Graves' Disease Study. J Thyroid Res. 2014;2014:165487. doi: 10.1155/2014/165487.
- Se-yeast 200 Microgr/day + arm A (Experimental): Additional arm where patients have been taking Se supplements during RISG1 therapy, and for 2 years after ATD withdrawal.
  Interventions: Other: Stop medication

INTERVENTIONS:
Other: Stop medication — Stop medication Stop medication + se supplement
  Other Names: stop medication + se supplement
  Arms: Se-yeast 200 Microgr/day + arm A; Stop of medication after remission

SUMMARY:
ATD therapy for Graves' disease is one of the commonly used options for therapy of the hyperthyroidism. The investigators study how to optimally keep patients in remission.

DETAILED DESCRIPTION:
A detailed description of patients entering the initial observational phase of the study (RISG1) has been published:

Laurberg P, Nygaard B, Andersen S, Carlé A, Karmisholt J, Krejbjerg A, Pedersen IB, Andersen SL. Association between TSH-Receptor Autoimmunity, Hyperthyroidism, Goitre, and Orbitopathy in 208 Patients Included in the Remission Induction and Sustenance in Graves' Disease Study. J Thyroid Res. 2014;2014:165487. doi: 10.1155/2014/165487.

ELIGIBILITY:
Inclusion Criteria:

* Graves hyperthyroidism in remission after ATD

Exclusion Criteria:

* Age < 18, severe concomitant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2008-01-07 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2015-05-15 (Actual)

PRIMARY OUTCOMES:
Relapse of hyperthyroidism | 2 years

SECONDARY OUTCOMES:
Reoccurrence of TSH-receptor autoimmunity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jesper S Karmisholt, MD, Ph.D, Principal Investigator — Aalborg University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karmisholt J, Andersen SL, Bulow-Pedersen I, Carle A, Krejbjerg A, Nygaard B. Predictors of Initial and Sustained Remission in Patients Treated with Antithyroid Drugs for Graves' Hyperthyroidism: The RISG Study. J Thyroid Res. 2019 Jan 3;2019:5945178. doi: 10.1155/2019/5945178. eCollection 2019. PMID 30719273